CLINICAL TRIAL: NCT06715124
Title: A Phase 1 Trial Evaluating the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Activity of QTX3544 in Patients With Advanced Solid Tumors With KRAS G12V Mutations
Brief Title: QTX3544 in Patients With Advanced Solid Tumors With KRAS G12V Mutations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Quanta Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QTX3544-201
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1a: QTX3544 monotherapy dose escalation (Experimental): QTX3544 will be administered at protocol defined dose based on cohort assignment
  Interventions: Drug: QTX3544
- Part 1b: QTX3544 dose escalation in combination with cetuximab (Experimental): QTX3544 will be administered at protocol defined dose in combination with cetuximab based on cohort assignment
  Interventions: Drug: QTX3544; Combination Product: Cetuximab
- Part 2: QTX3544 monotherapy dose expansion (Experimental): QTX3544 will be administered at protocol defined dose based on cohort assignment
  Interventions: Drug: QTX3544
- Part 3: QTX3544 dose expansion in combination with cetuximab (Experimental): QTX3544 will be administered at protocol defined dose in combination with cetuximab based on cohort assignment
  Interventions: Drug: QTX3544; Combination Product: Cetuximab

INTERVENTIONS:
Drug: QTX3544 — QTX3544 will be administered at protocol defined dose.
Combination Product: Cetuximab — Cetuximab will be administered at protocol defined dose.
  Arms: Part 1b: QTX3544 dose escalation in combination with cetuximab; Part 3: QTX3544 dose expansion in combination with cetuximab

SUMMARY:
Phase 1 study to determine the safety, tolerability, and anti-tumor activity of QTX3544 as a single agent or in combination with cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented, locally advanced or metastatic malignancy with KRAS G12V mutations identified through molecular testing (NGS- or PCR-based) with a Clinical Laboratory Improvement Amendments-certified (or equivalent) diagnostic.
* Part 1: Advanced solid tumors with at least one prior systemic therapy.
* Evaluable and measurable disease per RECIST v1.1.
* Part 2 and 3: Measurable disease per RECIST v1.1.

Exclusion Criteria:

* Active brain metastasis or carcinomatous meningitis
* Significant cardiovascular disease
* Active infection requiring intravenous (IV) antibiotics
* Prior treatment with a KRAS inhibitor

Other protocol-defined Inclusion/Exclusion Criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2027-01-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | up to 2 years
  Define as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug monotherapy and in combination with cetuximab.
Number of participants with Dose Limiting Toxicities (DLTs) | up to 21 days
  DLTs will be defined as the occurrence of any of the toxicities as described in the protocol.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of QTX3544 | up to 2 years
  Plasma concentration data for QTX3544 will be used to evaluate the area under the concentration-time curve (AUC) of QTX3544.
Peak plasma concentration of QTX3544 (Cmax) | up to 2 years
  Plasma concentration data for QTX3544 will be used to evaluate peak plasma concentration (Cmax) of QTX3544.
Objective response rate (ORR) | up to 2 years
  The ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) based on RECIST 1.1.
Duration of response (DoR) | up to 2 years
  DoR is defined as the time between first evidence of objective response and disease progression (as measured by RECIST 1.1) or death, whichever occurs earlier, in subjects who achieve CR or PR.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Sarah Cannon Research Institute, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - South Texas Accelerated Research Therapeutics, LLC Midwest, Grand Rapids, Michigan
  - Duke Cancer Center, Durham, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - South Texas Accelerated Research Therapeutics Mountain Region, LLC, West Valley City, Utah